CLINICAL TRIAL: NCT02467881
Title: Physical Activity and Sedentary Behavior Change; Impact on Lifestyle Intervention Effects for Diabetes Translation
Brief Title: Physical Activity and Sedentary Behavior Change; Impact on Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Kriska, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20050105; R18DK100933-02 (NIH)
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-02

CONDITIONS: Sedentary Lifestyle; Physical Activity
Keywords: Physical Activity; Sedentary; Lifestyle Intervention
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (3):
- Physical Activity Increase (GLB-MOD) (Active Comparator): Participants randomized to this arm will follow the traditional GLB program with an activity goal of 150 minutes per week of moderately intense physical activity similar to a brisk walk. Progression of the activity goal each week is slow and safe with increases of no more than 30 minutes per week. Participants are requested to try and achieve 20-30 minutes per day of moderate activity but, to allow for flexibility, that amount can be split into 10 minute increments. Self-reported monitoring for this group includes keeping track of weight, daily food intake as well the number of minutes each day spent being active as part of their planned activity goal. This is all recorded in the self-monitoring keeping track book.
  Interventions: Behavioral: Physical Activity Increase (GLB-MOD)
- Sedentary Time Decrease (GLB-SED) (Active Comparator): The GLB curriculum will be adapted to direct participants to decrease the time they spend sitting in a day rather than to increase moderate+ physical activity as is the case in the current GLB program. In order for the participant to become aware of how much time they spend sitting and where most of their sitting time occurs, they will fill out a "7 Day Sedentary Diary" that consists of daily entry of time spent sitting over the course of one week. Participants will be asked to eliminate a 45 minute sitting bout in a day with non-sitting activity. They will initially be asked to eliminate 45 minutes of sitting for two days in that week. This will increase one day a week until 7 days in a week are met.
  Interventions: Behavioral: Sedentary Time Decrease (GLB-SED)
- 6-month delayed (DELAYED) (Other): Those assigned to the DELAYED group at baseline will wait for 6 months to begin intervention. During the delayed time period, these participants will receive periodic health information newsletters. At the end of 6 months, the DELAYED participants will be randomly assigned to GLB-MOD or GLB-SED intervention, and will begin their intervention program at that time.
  Interventions: Other: 6-month delayed (DELAYED)

INTERVENTIONS:
Behavioral: Physical Activity Increase (GLB-MOD) — The Group Lifestyle Balance (GLB) program was adapted from the original DPP lifestyle intervention. As in the original DPP lifestyle program, the GLB goals are to achieve and maintain a 7% weight loss, and to safely and progressively increase physical activity to 150 minutes/week of moderately intense physical activity similar to a brisk walk.
  The curriculum will be administered in intervention groups with an average of 10-15 individuals per group; sessions will be conducted by trained coaches, with participants attending 22 sessions over one year.
  The two intervention arms will only differ in the aerobic activity portion of the intervention, which is covered in sessions #4, #10 and 19 as well as participant record keeping and goal setting in regards to activity/inactivity progression.
  Arms: Physical Activity Increase (GLB-MOD)
Behavioral: Sedentary Time Decrease (GLB-SED) — As in the original DPP, the GLB goal for weight is to achieve and maintain a 7% weight loss. For this intervention arm, instead of focusing on increasing moderate physical activity, the GLB curriculum will be adapted to address decreasing sitting time. Participants will have a goal of decreasing sitting time by 45 minutes/day. The curriculum will be administered in intervention groups with an average of 10-15 individuals per group; sessions will be conducted by trained coaches, with participants attending 22 sessions over one year.
  The two intervention arms will only differ in the aerobic activity portion of the intervention, which is covered in sessions #4, #10 and 19 as well as participant record keeping and goal setting in regards to activity/inactivity progression.
  Arms: Sedentary Time Decrease (GLB-SED)
Other: 6-month delayed (DELAYED) — Individuals assigned to 6 month delay will wait for 6 months from baseline to be randomly assigned to one of the two interventions and will begin intervention at that time. During the waiting period they will receive health information newsletters.
  Arms: 6-month delayed (DELAYED)

SUMMARY:
Diabetes Prevention Program translational efforts, such as the Group Lifestyle Balance Program (GLB), have been shown to be effective in reducing weight and modifying diabetes and CVD risk factors in a variety of diverse community settings. Although one of the two primary goals of these DPP translation programs focuses on increasing physical activity levels, few published DPP translation studies reported results on change in physical activity with only one study reporting activity levels from an objective measurement instrument. In order to completely understand the role that physical activity plays in making healthy lifestyle change, it is critical that we validate the impact of activity using a valid and reliable objective measure. In addition, current studies suggest that decreasing time spent sitting may have a positive health impact separate from the effects of participating in planned bouts of moderate intensity activity. Therefore, we propose to examine the impact of a modified version of the GLB program, which will focus on decreasing sedentary/sitting behaviors. The results of this project will provide information regarding best options for physical activity within lifestyle intervention programs, focusing both on verifying the current role of physical activity in lifestyle intervention using an objective measure and on examining an alternative intervention option for translation efforts.

DETAILED DESCRIPTION:
Translation efforts based upon the successful Diabetes Prevention Program (DPP) have shown that this behavioral lifestyle intervention model is effective in a variety of diverse community settings. Despite the fact that physical activity is a key part of the DPP lifestyle intervention as one of the two intervention goals, activity change in the DPP, and/or the resulting translation studies modeled after it, has not been adequately verified with an accurate objective measure. In addition, previous research has shown that, in many subgroups of the general population, moderate and vigorous physical activity is non-existent. Individuals with activity only at the low end of the intensity spectrum may have a difficult time increasing their levels of moderate+ intensity physical activity for various reasons such as limited function or lack of motivation. For these individuals, interventions with a movement goal of increasing planned bouts of moderate intensity activity may not be as effective and therefore not as beneficial as interventions with a movement goal of decreasing time spent sitting.

The purpose of this proposal is to understand the impact of movement, specifically physical activity and sitting time, in a DPP-adapted community lifestyle intervention, Group Lifestyle Balance (GLB).

Aim 1: To determine if the GLB lifestyle intervention, shown to be effective in translation efforts in decreasing weight and increasing self-reported activity, has significant changes in physical activity levels determined by a validated objective measure, the accelerometer. It is hypothesized that participants randomized to the conventional lifestyle intervention arm (GLB-MOD) will have significant improvements in our primary endpoints of weight and physical activity (measured objectively) compared to a delayed-intervention control at 6 months and will have reductions in several secondary outcome measures (fasting glucose, insulin, blood pressure, waist, lipids, physical function, and quality of life).

Aim 2: To determine if a lifestyle intervention program similar to the one described above, with the only change being that the activity focus is now replaced with an inactivity focus (GLB-SED), is also effective. It is hypothesized that participants randomized to GLB-SED will have a significant improvement in the primary endpoints of weight and decreased inactivity (measured objectively) compared to a delayed-intervention control at 6 months and will have significant reductions in several of the secondary endpoints (fasting glucose, insulin, blood pressure, waist circumference, lipids, physical function, quality of life).

Secondary Aims: To examine the pre-post change in participants for weight, physical activity (objective and subjective), and sedentary time from baseline to 6 and 12 months of intervention for each randomized arm and to understand the inter-relationships of these behavioral factors over time. It is hypothesized that those GLB-MOD participants who achieve significant weight loss will also have significant increases in their moderate+ intensity activity levels. Similarly, we hypothesize those GLB-SED participants who achieve significant weight loss will also have significant decreases in the amount of time they spent sedentary/sitting. An estimate of the difference in participant cost between the two versions of the lifestyle intervention programs will also be determined.

Aim #1 addresses an important remaining gap in the prevention literature; does objectively measured activity improve as a result of the existing intervention that is being used in DPP-based translation efforts and does this change in activity have an impact on weight change? Aim #2 examines the impact of replacing the conventional physical activity goal of increasing planned and relatively brief bouts of moderate physical activity with one focusing on decreasing sedentary time within the framework of a successful translation lifestyle intervention adapted from the DPP, the Group Lifestyle Balance (GLB) program.

The study design is a prospective, six month delayed-control intervention in which 321 subjects (age 50 and older with a BMI of ≥24 kg/m2 and with prediabetes and/or metabolic syndrome) will be recruited from community centers and randomly assigned to one of three groups: the standard GLB program which includes the conventional moderate activity goal (GLB-MOD), the GLB program with a focus on decreasing sedentary behavior (GLB-SED), or delayed intervention. Subjects assigned to GLB-MOD and GLB-SED will each, separately be compared at 6 months to the delayed-control group after which time, the delayed group will be randomly assigned to either GLB-MOD or GLB-SED. Participants will complete baseline, 6, and 12 month assessment visits. Change in weight, objectively measured activity, and time spent sedentary are the primary outcomes with secondary outcomes including change in self-reported physical activity, HbA1c, fasting glucose, lipids, blood pressure, waist circumference, quality of life and physical function.

It is hypothesized that physical activity assessed by accelerometry in GLB-MOD will significantly increase (mostly moderate intense activity) and that there will be a significant decrease in weight, which will partly be related to change in activity levels. The 2nd hypothesis is that the GLB-SED intervention will significantly decrease time spent sitting as measured by accelerometry and that this change will also be related to a significant decrease in weight. The information that will be gained from this entire effort is important, innovative, and will allow us to obtain a complete and accurate understanding of both ends of the physical activity/inactivity spectrum and their impact in community prevention intervention programs. If shown to be effective, the innovative, modified sedentary-focused translation intervention program would provide a valuable future translation option.

ELIGIBILITY:
Inclusion Criteria:

Individuals attending screening who are found to have prediabetes AND/OR the metabolic syndrome are eligible to participate in the intervention. Pre-diabetes is defined as having a fasting glucose >100 mg/dL and <126mg/dL and/or a hemoglobin A1C of 5.7%-6.4%.

Metabolic syndrome is defined as having at least 3 of the 5 following risk factors:

1. Waist circumference (>40 inches men, >35 inches women);
2. Blood pressure >130 mmHg (systolic) or >85 mmHg (diastolic) OR history of diagnosed hypertension
3. Low HDL level (<40mg/dL men, <50 mg/dL women)
4. Elevated triglyceride level >150 mg/dL
5. Fasting glucose >100mg/dL and <126mg/dL

Individuals attending screening with hyperlipidemia plus one additional component of the metabolic syndrome are also eligible.

Exclusion Criteria:

Individuals who are identified as having diabetes as a result of the screening are not eligible. All individuals enrolled in the study should have at least 6th grade English reading/writing ability. Physician approval will be requested to clear for the activity portion of the program.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
BMI (Body Mass Index) | Change in BMI between Baseline and 6 months
  BMI will be calculated as average weight divided by average height squared (kg/m2).
BMI (Body Mass Index) | Change in BMI between Baseline and 12 months
  BMI will be calculated as average weight divided by average height squared (kg/m2).
Actigraph Accelerometry | Change in Physical Activity Level between Baseline and 6 months
  Physical activity level objectively measured using Actigraph Accelerometry. This will be worn on the waist and will passively record physical activity and sedentary behavior.
Actigraph Accelerometry | Change in Physical Activity Level between Baseline and 12 months
  Physical activity level objectively measured using Actigraph Accelerometry. This will be worn on the waist and will passively record physical activity and sedentary behavior.

SECONDARY OUTCOMES:
Gait Speed | Change in Gait Speed between Baseline and 6 months
  Gait Speed (m/s over 4 m) will be used to measure change in physical function.
Gait Speed | Change in Gait Speed between Baseline and 12 months
  Gait Speed (m/s over 4 m) will be used to measure change in physical function.
Fasting glucose test | Change in Fasting glucose between Baseline and 6 months
  Blood sample
Fasting glucose test | Change in Fasting glucose between Baseline and 12 months
  Blood sample
Fasting lipid profile test | Change in Fasting lipid profile between Baseline and 6 months
  Blood sample
Fasting lipid profile test | Change in Fasting lipid profile between Baseline and 12 months
  Blood sample
Fasting Insulin test | Change in Fasting Insulin between Baseline and 6 months
  Blood test
Fasting Insulin test | Change in Fasting Insulin between Baseline and 12 months
  Blood test
Hemoglobin A1c test | Change in Hemoglobin A1c between Baseline an 6 months
  Blood sample
Hemoglobin A1c test | Change in Hemoglobin A1c between Baseline and 12 months
  Blood sample
Blood pressure | Change in Blood Pressure between Baseline and 6 months
Blood pressure | Change in Blood Pressure between Baseline and 12 months
Modifiable Activity Questionnaire | Change in self-reported Modifiable Activity Questionnaire between Baseline and 6 months
  The Modified Activity Questionnaire is a self-report of physical activity level and sedentary behavior.
Modifiable Activity Questionnaire | Change in self-reported Modifiable Activity Questionnaire between Baseline and 12 months
  The Modified Activity Questionnaire is a self-report of physical activity level and sedentary behavior.
EQ-5D Quality of Life Survey | Change in Quality of Life between Baseline and 6 months
  The EQ-5D quality of life survey measures health status and outcomes.
EQ-5D Quality of Life Survey | Change in Quality of Life between Baseline and 12 months
  The EQ-5D quality of life survey measures health status and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Kriska, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Epidemiology Department, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ratner R, Goldberg R, Haffner S, Marcovina S, Orchard T, Fowler S, Temprosa M; Diabetes Prevention Program Research Group. Impact of intensive lifestyle and metformin therapy on cardiovascular disease risk factors in the diabetes prevention program. Diabetes Care. 2005 Apr;28(4):888-94. doi: 10.2337/diacare.28.4.888. PMID 15793191
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Orchard TJ, Temprosa M, Goldberg R, Haffner S, Ratner R, Marcovina S, Fowler S; Diabetes Prevention Program Research Group. The effect of metformin and intensive lifestyle intervention on the metabolic syndrome: the Diabetes Prevention Program randomized trial. Ann Intern Med. 2005 Apr 19;142(8):611-9. doi: 10.7326/0003-4819-142-8-200504190-00009. PMID 15838067
- [Background] Kramer MK, Kriska AM, Venditti EM, Miller RG, Brooks MM, Burke LE, Siminerio LM, Solano FX, Orchard TJ. Translating the Diabetes Prevention Program: a comprehensive model for prevention training and program delivery. Am J Prev Med. 2009 Dec;37(6):505-11. doi: 10.1016/j.amepre.2009.07.020. PMID 19944916
- [Background] Kriska AM, Edelstein SL, Hamman RF, Otto A, Bray GA, Mayer-Davis EJ, Wing RR, Horton ES, Haffner SM, Regensteiner JG. Physical activity in individuals at risk for diabetes: Diabetes Prevention Program. Med Sci Sports Exerc. 2006 May;38(5):826-32. doi: 10.1249/01.mss.0000218138.91812.f9. PMID 16672833
- [Background] Wilmot EG, Davies MJ, Edwardson CL, Gorely T, Khunti K, Nimmo M, Yates T, Biddle SJ. Rationale and study design for a randomised controlled trial to reduce sedentary time in adults at risk of type 2 diabetes mellitus: project stand (Sedentary Time ANd diabetes). BMC Public Health. 2011 Dec 8;11:908. doi: 10.1186/1471-2458-11-908. PMID 22151909
- [Background] Steeves JA, Bassett DR, Fitzhugh EC, Raynor HA, Thompson DL. Can sedentary behavior be made more active? A randomized pilot study of TV commercial stepping versus walking. Int J Behav Nutr Phys Act. 2012 Aug 6;9:95. doi: 10.1186/1479-5868-9-95. PMID 22866941
- [Derived] Devaraj SM, Napoleone JM, Miller RG, Rockette-Wagner B, Arena VC, Mitchell-Miland C, Saad MB, Kriska AM. The role of Sociodemographic factors on goal achievement in a community-based diabetes prevention program behavioral lifestyle intervention. BMC Public Health. 2021 Oct 2;21(1):1783. doi: 10.1186/s12889-021-11844-z. PMID 34600527
- See also: Diabetes Prevention Support Center of the University of Pittsburgh — http://www.diabetesprevention.pitt.edu